CLINICAL TRIAL: NCT00685451
Title: Cognitive Therapy for PTSD in Addiction Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Mark P. McGovern, Ph.D., Principal Investigator, Dartmouth Medical School
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5K23DA016574 (NIH); 5K23DA016574 (NIH)
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2011-09-29 (Estimated); Status verified 2011-09

CONDITIONS: Stress Disorders, Post Traumatic; Substance-Related Disorders
Keywords: cognitive behavior therapy; addiction; PTSD
MeSH Terms: conditions — Combat Disorders; Substance-Related Disorders; Behavior, Addictive; Stress Disorders, Post-Traumatic | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT)

SUMMARY:
The purpose of this phase of the study is to assess the feasibility of a cognitive behavioral therapy for post-traumatic stress disorder (PTSD) in persons receiving outpatient services at an addiction treatment program. The next phase of the study will be a more rigorous investigation of the efficacy of the PTSD therapy within addiction treatment settings.

DETAILED DESCRIPTION:
PTSD is a common co-occurring disorder with substance use disorders (SUDs). When present, PTSD causes more negative outcomes in treatments designed to address substance use disorders. These negative outcomes include: 1) Early drop-out from treatment; 2) More frequent relapse to alcohol and other drugs; 3) Greater difficulty utilizing group therapies and self-help recovery groups; 4) Worsening of PTSD symptoms; and 5) Addiction treatment clinician distress. Nonetheless, the traditional practice in addiction treatment programs has been to address the problems of addiction, and delay treatment for PTSD and other psychiatric conditions. The evidence for negative outcomes for persons with co-occurring PTSD and SUDs challenges this practice, and suggests the need for new intervention strategies. A promising intervention for PTSD has emerged in another at-risk and vulnerable population of persons already receiving treatment for their "primary" disorder. This is a cognitive behavioral therapy for PTSD in persons with severe mental illness (SMI). Pilot studies with this intervention have demonstrated effectiveness, that it is well tolerated by patients, and that it fits within existing treatment services. Given the high prevalence of co-occurring PTSD and SUDs in addiction treatment settings (33-59%), the negative outcomes associated with this comorbidity, and the potential availability of a promising intervention, a stage one feasibility study appears warranted.

Patients admitted to an addiction treatment program are routinely screened for PTSD using a brief self-report survey, the PTSD Checklist (PCL). These forms are collected by clinical staff of the treatment program and scored for PTSD diagnostic criteria. If a patient exceeds threshold criteria (PCL score of greater than or equal to 44) they are approached by a clinical staff member about their potential interest in the study. If they wish to learn more about the study the PI or designee is contacted, a suitable time arranged, and the patient approached for their interest in consenting to the study.

If consent is granted, the subject is interviewed by a member of the research team and demographic, substance use, and treatment history information is extracted from the subject's medical record. The interview consists of standardized procedures (Clinician Administered PTSD Scale [CAPS], SCID-Axis II borderline personality disorder) designed to assess PTSD and other commonly associated psychiatric disorders. A urine screen and breathalyzer are conducted to test for alcohol and other drugs. Self-report measures of depression (Beck Depression Inventory-II [BDI-II]), anxiety (Beck Anxiety Inventory [BAI]), alcohol and drug use (Addiction Severity Index [ASI] and Time-line Follow-back Calendar), treatment readiness for substance use (Stages of Change Readiness and Treatment Eagerness Scale [SOCRATES]) and for PTSD (SOC-PTSD), HIV risk (HIV-risk Screening Instrument [HSI]), and treatment utilization (Recent Treatment Survey [RTS]) are also administered. If the subject again meets criteria for PTSD (CAPS confirms diagnosis of DSM-IV PTSD), he or she is presented with the opportunity to receive the PTSD cognitive behavioral therapy. In either case, the subject receives $25 for participating in the interview.

The cognitive behavioral therapy is conducted in individual sessions, approximately 50 minutes in duration. The therapy is manual-guided, focused on the PTSD symptoms only, and designed to work in conjunction with the addiction treatment program services. The therapy is offered in weekly sessions, for 12-14 total sessions. At monthly intervals, the subject will complete the RTS and a trauma event checklist based on the PCL, and will be tested for alcohol (breathalyzer) and drug use (urine screen). The subject will also complete the Working Alliance Inventory (WAI - client version) after the second PTSD therapy session.

At completion of the PTSD therapy the patient will again be interviewed by a member of the research team. The post-therapy assessment will consist of the CAPS, the Time-line Follow-back, BAI, BDI-II, RTS, ASI, HSI, and a measure of treatment satisfaction (Client Satisfaction Questionnaire [CSQ-8]). The subject is again compensated $25 for the post-therapy assessment. At three months post completion, the subject participates in a follow-up interview. This interview will consist of the same measures used at the post-therapy assessment, with the exception of the CSQ-8 and with the addition of the trauma event checklist. The subject is again compensated $25 for their participation in the follow-up interview. All research activities, including all assessments and therapy sessions, will be conducted on-site at the addiction treatment program.

We plan to enroll approximately 100 subjects in the feasibility phase of the study. The subject outcome and program experiences with the protocol will be used in planning the subsequent pilot trial phase of the study. The pilot trial will be a larger, randomized controlled trial comparing the study cognitive behavioral therapy with a matched-attention control condition.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old;
* Actively enrolled in intensive outpatient addiction services;
* Diagnosis of PTSD; and
* Willing and able to provide informed consent.

Exclusion Criteria:

* Acute psychotic disorder;
* Psychiatric hospitalization or suicide attempt in the past 2 months;
* Known impending court appearance or legal circumstance that may result in incarceration within next 8 months; and
* Known medical condition that would likely cause study withdrawal in the next 8 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2004-11; Primary Completion 2006-08 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
decrease in substance use at post-therapy and 3 month follow-up
reduction in PTSD symptoms at post-therapy and 3 month follow-up
improvement in addiction treatment retention

SECONDARY OUTCOMES:
examine impact of depression, anxiety, and borderline personality disorder on outcomes
explore impact of motivation and treatment readiness on outcomes
assess overall level of satisfaction with treatment on outcomes
examine impact of other services received on outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Mark P. McGovern, Ph.D., Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (3):
- United States (3):
  - Fresh Start at Concord Hospital, Concord, New Hampshire
  - Farnum Center, Manchester, New Hampshire
  - Quitting Time, Wilder, Vermont